CLINICAL TRIAL: NCT05813314
Title: A Phase 1, Randomized, Open-Label, Sponsor-Open, Two-Sequence, Two-Period Crossover Study to Investigate the Bioequivalence of a Single Subcutaneous Dose of BMN 111 Administered Using Either a Vial and Syringe or Injector Pen in Healthy Adult Participants
Brief Title: Bioequivalence Study to Compare Two Injection Devices for BMN 111 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The BMN 111-104 study has terminated as further optimization of the approach to achieve bio equivalence is required. The study termination was not due to any patient safety concerns.
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 111-104
Record Dates: First submitted 2023-03-16; First posted 2023-04-14 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia | interventions — Syringes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BMN 111 injection with vial and syringe (Active Comparator): Study treatment will be provided in glass vials. Each glass vial will be labeled as required per country requirement. Pre-filled Diluent Transfer Syringes will be provided for reconstitution.
  Interventions: Drug: BMN 111 administration via vial and syringe
- BMN 111 injection with injector pen (Experimental): Study treatment will be provided in a prefilled injector pen containing a dual chamber drug cartridge, for reconstitution and injection, after setting of the specified dose with the 2.0 mg/mL formulation.
  Interventions: Combination Product: BMN 111 administration via Injector Pen

INTERVENTIONS:
Combination Product: BMN 111 administration via Injector Pen — BMN 111 Injection will be given using an injector pen
  Arms: BMN 111 injection with injector pen
Drug: BMN 111 administration via vial and syringe — BMN 111 Injection will be given using vial and syringe
  Arms: BMN 111 injection with vial and syringe

SUMMARY:
The purpose of this study is to establish the bioequivalence of a single SC dose of BMN 111 administered using a vial and syringe versus using an injector pen.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged 18 to 55 years inclusive, at the time of signing the informed consent.
2. Participants must be non-smoking (have never smoked, or stopped smoking > 3 months prior to dosing), and can be of any ethnicity.
3. Participants must be healthy as determined by the absence of clinically relevant abnormalities identified by medical evaluation, including medical history, full physical examination, laboratory tests, cardiac monitoring, supine vital signs to include temperature, and assessment of prior and concomitant medications.
4. Body weight ≥ 60 kg and < 110 kg and body mass index within the range 18.0 to 32.0 kg/m2 (inclusive).
5. Males and/or females are eligible to participate in this clinical study.
6. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
7. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
8. Participants must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria:

1. Any condition considered to affect drug absorption (eg, conditions affecting SC administration such as reduced SC blood flow, lipohypertrophy, and significantly high/low skin temperature).
2. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
4. History of migraines.
5. Confirmed (eg, two consecutive measurements) systolic blood pressure > 140 or < 90 mmHg, diastolic blood pressure > 90 or < 50 mmHg, and pulse rate > 100 or < 40 beats per minute or recurrent symptomatic hypotension (defined as episodes of low BP generally accompanied by symptoms e.g., dizziness and fainting) or recurrent symptomatic orthostatic hypotension.
6. Positive hepatitis panel and/or positive human immunodeficiency virus test.
7. Exposure to mycobacterium tuberculosis, indicative of tuberculosis infection, as confirmed by a positive QuantiFERON-TB Gold test.
8. A positive COVID-19 test at Screening or Check-in.
9. Taking any of the prohibited medications.
10. Administration of a coronavirus disease 2019 (COVID-19) vaccine within 30 days prior to dosing.
11. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the investigator (or designee).
12. Use or intend to use any prescription medications/products other than hormone replacement therapy (HRT), oral, implantable, transdermal, injectable, or intrauterine contraceptives within 7 days (or 14 days if the drug is a potential enzyme inducer), or 5 half-lives (whichever is longer), prior to dosing, unless deemed acceptable by the investigator (or designee).
13. Use or intend to use slow release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the investigator (or designee).
14. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days, or 5 half-lives (whichever is longer), prior to dosing, unless deemed acceptable by the investigator (or designee).
15. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives prior to dosing (whichever is longer).
16. Have previously completed or withdrawn from this study or any other study investigating BMN 111 and have previously received BMN 111.
17. Aspartate aminotransferase, alanine aminotransferase, or bilirubin ≥ 1.5 × upper limit of normal or estimated glomerular filtration rate < 60 mL/min/1.73m2 (Chronic Kidney Disease Epidemiology Collaboration 2021).
18. Receipt of blood products within 2 months prior to Check-in.
19. Donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
20. Poor peripheral venous access.
21. Participants who, in the opinion of the investigator (or designee), should not participate in this study.
22. Any skin condition, such as scarring or tattoos, which may preclude receipt of the study drug.
23. Unwilling or unable to comply with scheduled visits, the treatment plan, laboratory tests and other study procedures or lifestyle guidance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration (Cmax) | Predose, 2, 5, 15, 30, 45, 60, and 75 minutes and 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose
Area under the concentration versus time curve from time 0 to infinity (AUC0-∞) | Predose, 2, 5, 15, 30, 45, 60, and 75 minutes and 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose
Area under the concentration versus time curve from time 0 to t, where t is the last timepoint with a measurable concentration (AUC0-t) | Predose, 2, 5, 15, 30, 45, 60, and 75 minutes and 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose

SECONDARY OUTCOMES:
Time of Cmax (tmax) | Predose, 2, 5, 15, 30, 45, 60, and 75 minutes and 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose
Time of t1/2 | Predose, 2, 5, 15, 30, 45, 60, and 75 minutes and 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose
Time of terminal rate constant (λZ) | Predose, 2, 5, 15, 30, 45, 60, and 75 minutes and 1.5, 2, 2.5, 3, 4, 6, and 8 hours postdose
Incidence and severity of adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp, Dallas, Texas, United States